CLINICAL TRIAL: NCT02768662
Title: A 6-Month, Multicenter, Phase 3, Open-Label Extension Safety Study of OTO-104 Given At 3-Month Intervals by Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: A 6-Month Extension Study of OTO-104 in Meniere's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Negative Efficacy Results from the recently completed Phase 3 study 104-201506
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-201610
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTO-104 (Experimental): 12 mg dexamethasone
  Interventions: Drug: OTO-104

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg OTO-104

SUMMARY:
This is an open-label extension study of a single intratympanic injection of OTO-104 given every 3 months for a total of 2 injections. Subjects must have completed either Otonomy study 104-201403 (1-Year, Phase 2, Safety Study of OTO-104) or 104-201508 (Phase 3 Study of OTO-104) in order to be eligible for this open-label extension study.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has completed the Phase 2 OTO-104 1-Year Safety Study (104-201403) or Phase 3 (104-201508) clinical study.
* Subject has a diagnosis of definite unilateral Meniere's disease by 1995 AAO-HNS criteria

Exclusion Criteria includes, but is not limited to:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has experienced an adverse reaction to intratympanic injection of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Many sites in Europe. Refer to the contact info listed below., San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 142 subjects were enrolled. Of the 142 subjects enrolled, 46 had previously completed the 104-201403 study and 96 had previously completed the 104 201508 study. The first subject enrolled on August 25, 2016, and the last subject completed on September 8, 2017.
Pre-assignment Details: This study was terminated early based on results of study 104-201506, a US Phase 3 study that indicated no statistically significant difference in the primary endpoint of reduction in definitive vertigo days (DVD) for OTO-104 vs placebo nor for any of the secondary endpoints. Decision was made to terminate all ongoing studies on August 31, 2017, including this study. At the time of termination, 90 subjects completed the study through Month 3 and 56 subjects completed the study through Month 6.
Groups:
- OTO-104: Intratympanic injection of 12 mg OTO-104
Period: Overall Study
Arm/Group | OTO-104
Started | 142
Completed | 56
Not Completed | 86
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 3
Not completed — Study terminated by Sponsor | 78

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Groups:
- OTO-104: 12 mg dexamethasone
  OTO-104: Intratympanic injection of 12 mg OTO-104
Arm/Group | OTO-104
Number analyzed (Participants) | 142
Age, Continuous [Median (Full Range); unit: years] | 53.0 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 136
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Belgium | 6
  France | 4
  Germany | 17
  Italy | 9
  Poland | 23
  United Kingdom | 83
Duration of Meniere's Disease [Count of Participants; unit: Participants]
  ≤5 years | 109
  6-10 years | 18
  11-15 years | 8
  >15 years | 7

OUTCOME MEASURES:

1. Primary Outcome: Otoscopic Examination - Tympanic Membrane Perforation at Week 24 (Month 6)
Description: Otoscopic exams were conducted at each visit. It was considered important to understand if the tympanic membrane perforation that resulted from the IT injection persisted at the end of study visit (24 Weeks [Month 6]).
Time Frame: 6 Months
Population: The 6-month Safety Analysis Set included all subjects who received at least 1 dose of study drug and completed the Month 6 visit
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104
Number analyzed (Participants) | 56
Participants
  Perforation present: pinhole size | 0
  Perforation present: ≤25% tympanic membrane | 0
  Perforation present: >25% and ≤50% tympanic membrane | 0
  Perforation present: >50% tympanic membrane | 0
  Perforation not present | 56
  Perforation information missing | 0

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug up until the end of the study (Month 6).
Arm/Group | OTO-104
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 4/142
Other Adverse Events (participants affected / at risk) | 37/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=142)
Abdominal Pain and Constipation (Gastrointestinal disorders) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=142)
Nasopharyngitis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 4 (4)
Meniere's Disease (Ear and labyrinth disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Injection Site Discomfort (General disorders) | 3 (3)
Procedural Dizziness (Injury, poisoning and procedural complications) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02768662/Prot_SAP_000.pdf